CLINICAL TRIAL: NCT06126458
Title: Okçuluk Sporcularında Stabilizasyonun ve Stabilizasyonla İlişkili Parametrelerin Atış Performansına Olan Etkisinin Servikal, Lumbal ve Skapular Seviyede İncelenmesi
Brief Title: the Effect of Stabilization on Archery Performance
Status: Completed | Type: Observational
Sponsor: Aynur Demirel (Other)
Responsible Party: Sponsor-Investigator, Aynur Demirel, PT, PhD, Assoc. Prof., Hacettepe University
Organization: Hacettepe University (Other)
Other Study IDs: GO21/1028
Record Dates: First submitted 2023-01-30; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Athletic Injuries; Instability, Joint
MeSH Terms: conditions — Athletic Injuries; Joint Instability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Good shooting performance: archery athletes who had 589 and more
  Interventions: Other: shooting performance
- Bad shooting performance: archery athletes who had 588 and less
  Interventions: Other: shooting performance

INTERVENTIONS:
Other: shooting performance — collecting total points after 72 target shootings done

SUMMARY:
The aim of this study was to investigate the effect of stabilization and stabilization-related parameters on shooting performance at the cervical, lumbal and scapular levels in archery athletes. A total of 40 archery athletes aged between 10 and 18, who have been professionally engaged in archery for at least 1 year were included in the study. Demographic information and musculoskeletal system evaluations of the athletes were done. Performance of the athletes via Upper Extremity Closed Kinetic Chain Stability Test, Hand Grip Strength test; presence of scapular dyskinesia was evaluated via the Lateral Scapular Slide Test. Cervical region stabilization was evaluated via Craniocervical Flexion Test, scapular level stabilization was evaluated via Scapular Muscle Endurance Test, lumbar region stabilization was evaluated via Abdominal Drawing-in Test and Sahrmann's Core Stability Test. As the parameters related to stabilization, postures via Corbin Postural Rating Scale; balances via Stork Balance Test, Upper Extremity Y Balance Test; pain was evaluated via the Shoulder Pain and Disability Index. Shooting performances were evaluated with 72 target shootings and a total of 720 points. .

DETAILED DESCRIPTION:
Archery can be described as a comparatively static sport requiring strength and endurance of the upper body, in particular the forearm and shoulder girdle. Skill in archery is defined as the ability to shoot an arrow to a given target in a certain time span with accuracy. The discipline is described as a three-phase (the stance, the drawing and the sighting) movement. Shooting can be divided these phases into six: bow hold, drawing, full draw, aiming, release and follow-through. Each of these phases represented a stable sequence of movements and was ideal for studying the motor control and skill acquired during this voluntary kinematic process.

An archer pushes the bow with an extended arm, which is statically held in the direction of the target, while the other arm exerts a dynamic pulling of the bowstring from the beginning of the drawing phase, until the release is dynamically executed. The release phase must be well balanced and highly reproducible to achieve commendable results in a competition.

The bowstring is released when an audible impulse is received from a device called "clicker" that is used as a draw length check. Each arrow can be drawn to an exact distance and a standard release can be obtained using the device. The clicker is reputed to improve the archer's score and used by all target archers. The archer should react to the clicker as quickly as possible. In particular, a repeated contraction and relaxation strategy in the forearm and pull finger muscles should be developed for this reason.

The aim of this study was to investigate the effect of stabilization and stabilization-related parameters on shooting performance at the cervical, lumbal and scapular levels in archery athletes. A total of 40 archery athletes aged between 10 and 18, who have been professionally engaged in archery for at least 1 year were included in the study. Demographic information and musculoskeletal system evaluations of the athletes were done. Performance of the athletes via Upper Extremity Closed Kinetic Chain Stability Test, Hand Grip Strength test; presence of scapular dyskinesia was evaluated via the Lateral Scapular Slide Test. Cervical region stabilization was evaluated via Craniocervical Flexion Test, scapular level stabilization was evaluated via Scapular Muscle Endurance Test, lumbar region stabilization was evaluated via Abdominal Drawing-in Test and Sahrmann's Core Stability Test. As the parameters related to stabilization, postures via Corbin Postural Rating Scale; balances via Stork Balance Test, Upper Extremity Y Balance Test; pain was evaluated via the Shoulder Pain and Disability Index. Shooting performances were evaluated with 72 target shootings and a total of 720 points. .

ELIGIBILITY:
Inclusion Criteria:

* healty athletes who have been professionally engaged in archery for at least 1 year
* using same type of equipment(compound or recurve)
* being volunteer

Exclusion Criteria:

* who have orthopedic or neurological problems in last one year
* having structural or functional scoliosis
* no surgical operations
* BMI>30 kg/m2

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: healty elite archery athletes
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-11-06 (Actual); Study Completion 2022-11-06 (Actual)

PRIMARY OUTCOMES:
cervical stabilization | baseline
  cervical stabilization assess with craniocervical flexion test.
lumbar stabilization grade | baseline
  lumbar stabilization asses with sahrmann's core stability test and will grade according to test outcome.
lumbar stabilizator muscle contraction | baseline
  the athlete perform abdominal drawing in meneuver and contraction amount record.
scapular dyskinesis type | baseline
  Kibler's scapular diskinesis test and lateral scapular slide test
scapular dyskinesis amount | baseline
  lateral scapular slide test
sportive performance | baseline
  the athlete will shoot 72 arrows to the target and tthe total points will record as score.

SECONDARY OUTCOMES:
balance assessment | baseline
  upper extremity Y balance test
static balance assessment | baseline
  stand stork test
posture | baseline
  Corbin posture assessment
disability | baseline
  shoulder pain related disability will assess with The Shoulder Pain and Disability Index (SPADI). The SPADI has 13 items. Each item is scored on a visual analog scale (VAS) from 0 to 10, with 0 indicating no pain or no disability and 10 indicating the worst pain or disability possible. The total score ranges from 0 to 100, with higher scores indicating more pain and disability.
upper extremity performance | baseline
  upper extremity erformance assess with upper extremity closed chain stability test
hand grip strenght | baseline
  hand grip streng assess with hand dynamometer
muscle tightness | baseline
  pectoralis minor, shoulder abductor&internal rotator and trapezious muscle tightness assess

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Demirel, Assoc. Prof., Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Sıhhiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] 1. Book 3, Target Archery [Erişim Tarihi 18 Mayıs 2022]. Available from: https://rulebook.worldarchery.sport/PDF/Official/2021-01-01/EN-Book3.pdf 2. Target Archery [Erişim Tarihi 18 Mayıs 2022] [Available from: https://worldarchery.sport/sport/disciplines/target-archery. 3. Yönal G, Turkmen M. TÜRK KÜLTÜR YAŞAMINDA OKÇULUK. ASOS Journal. 2017;5:523-33. 4. Atabeyoğlu C. Okçuluk Tarihi. Ankara: Türk Spor Vakfı Yayınları Başkent Yayınevi; 1988. 5. Martin PE, Siler WL, Hoffman D. Electromyographic analysis of bow string release in highly skilled archers. Journal of Sports Sciences. 1990;8(3):215-21. 6. akınoğlu B, Kocahan T, Birben Kurt T, Çoban Ö, Soylu C, Yildirim N. Paralimpik Okçuların ve Tekerlekli Sandalye Basketbol Oyuncularının Core Stabilizasyon Verilerinin Karşılaştırılması. Online Türk Sağlık Bilimleri Dergisi. 2016;1:21-7. 7. History. [Erişim Tarihi 15 Mayıs 2022] [Available from: https://worldarchery.sport/sport/history. 8. Members. [Erişim Tarihi 15 Mayıs 2022] [Available from: https://worldarchery.sport/members. 9. Gazoz M, Şimşek Y. Okçuluk Ders Kitabı. Ankara: Milli Eğitim Bakanlığı Yayınları; 2019. 10. Indoor Archery [Erişim Tarihi 18 Mayıs 2022] [Available from: https://worldarchery.sport/sport/disciplines/indoor-archery. 11. Okçuluk-Yarışma-Talimatı V-01. [Erişim Tarihi 18 Mayıs 2022] [Available from: https://www.tof.gov.tr/federasyon/talimatlar/. 12. Equipment Erişim Tarihi 14 Mayıs 2022 [Available from: https://worldarchery.sport/sport/equipment. 13. Mohamed M, Azhar A. Postural Sway And Shooting Accuracy Of Skilled Recurve Archers. Movement, Health & Exercise. 2012;1. 14. Nishizono H, Shibayama H, Izuta T, Saito K. Analysis of Archery Shooting Techniques by Means of Electromyography. 1987. 15. Tak K-H. Archery: Korea Archery Association; 2012. 301 p. 16. Charles D. Archery: Skills. Tactics. Techniques: T.H.E. Crowood Press LTD; 2015. 17. Sarro K, Viana T, Barros R. Relationship between bow stability and postural control in recurve archery. European Journal of Sport Science. 2020;21. 18. Stone RT. The Biomechanical and Physiological link between Archery Techniques and Performance. Proceedings of the Human Factors and Ergonomics Society Annual Meeting. 2007;51(18):1227-31. 19. Spratford W, Campbell R. Postural stability, clicker reaction time and bow draw force predict performance in elite recurve archery. European Journal of Sport Science. 2017;17(5):539-45. 20. Shinohara H. Analysis of muscular activity in archery: A compar. 2018. 21. Vendrame E, Belluscio V, Truppa L, Rum L, Lazich A, Bergamini E, et al. Performance assessment in archery: a systematic review. Sports Biomechanics. 2022:1-23. 22. Lin J-J, Hung C-J, Yang C-C, Chen H-Y, Chou F-C, Lu T-W. Activation and tremor of the shoulder muscles to the demands of an archery task. Journal of sports sciences. 2010;28(4):415-21. 23. Azhar S, Sharma S, Sharma S, Tanwar T. EMG activity of transversus abdominis, multifidus and co-contraction index in different phases amongst varied level archers: A cross-sectional study. Polish Journal of Sport and Tourism. 2021;28(1):19-23. 24. Stone RT, editor The biomechanical and physiological link between archery techniques and performance. Proceedings of the human factors and ergonomics society annual meeting; 2007: SAGE Publications Sage CA: Los Angeles, CA. 25. Ahmad Z, Taha Z, Hassan HA, Hisham MA, Johari NH, Kadirgama K, editors. Biomechanics measurements in archery. International Conference on Mechanical Engineering Research (ICMER2013); 2013.